CLINICAL TRIAL: NCT03991026
Title: Farm to Clinic Vegetable Initiative at East Baltimore Medical Center
Brief Title: Healthy Foods and Education to Treat Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00164545
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of 2 groups: a control group or the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy food and Education/Cooking Classes (Experimental): At consent, participant will complete the baseline survey. Baseline survey will collect information like vegetable consumption, healthy eating attitudes, and demographics. Every week for 6 weeks, participants will pick-up a healthy food bag (e.g. fresh vegetables) for a $3 co-pay and attend an hour-long education classes at East Baltimore Medical Center. All participants will complete a survey at healthy food bag pick-up or an education class. Surveys at bag pick-up will ascertain outcomes like vegetable consumption. Surveys at education classes will ascertain outcomes like healthy eating attitudes. At 6 weeks, all participants will complete a follow-up survey equivalent to the baseline survey. The follow-up survey will be completed again at 10 weeks, 18 weeks, and 30 weeks. Participants will also be weighed at each bag pick-up (participants may decline) and relevant health information like blood pressure will be obtained from the EMR from an associated office visit.
  Interventions: Behavioral: Healthy food and Education/Cooking Classes
- Control Group (No Intervention): At consent, participant will complete the baseline survey. Baseline survey will collect information like vegetable consumption, cooking habits, food security, healthy eating attitudes, and demographics. As a control group, participants will not partake in the healthy food bag pick-ups or cooking classes therefore they will not fill out those associated surveys. After the 6 weeks of the intervention, control participants will be given the follow-up survey equivalent to the baseline survey. The follow-up survey will be completed again after 10 weeks, 18 weeks, and 30 weeks. Participants will also be weighed at each bag pick-up (participants may decline) and relevant health information like blood pressure will be obtained from the EMR from an associated office visit.

INTERVENTIONS:
Behavioral: Healthy food and Education/Cooking Classes — The intervention includes providing weekly seasonal produce and healthy foods to participants in addition to an education/cooking class that will be tailored to Diabetes Mellitus, Type II.
  Arms: Healthy food and Education/Cooking Classes

SUMMARY:
The investigators will study a program that delivers weekly community-supported agriculture shares to patients of East Baltimore Medical Center in order to increase access to healthy foods. The investigators will provide adult patients with uncontrolled diabetes with healthy foods including fresh vegetables and shelf-stable pantry items (e.g., canned beans) every week over the course of 6 weeks. The investigators will also collect demographic data and food insecurity status of participants via survey. This program will also conduct weekly cooking and nutrition classes at East Baltimore Medical Center. The investigators will conduct a survey of participants' experiences each time participants pick up a vegetable bag and at the end of the cooking classes. In addition, a focus group of participants will be held to gather qualitative data regarding the vegetable initiative.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uncontrolled diabetes mellitus (defined as a glycosylated hemoglobin >8%)
* 18 years age of and over
* Living within the geographical region of East Baltimore Medical Campus

Exclusion Criteria:

* Current participation in Five Plus Nuts and Beans Study or other program that provides diet-based food
* Non-English speaking
* On hospice or palliative care
* Acute or chronic psychosis
* Active substance or alcohol use disorder
* Another active medical disorder that would preclude participation in weekly food pick-up or classes including: active treatment of cancer, steroid dependent asthma/chronic obstructive pulmonary disease/emphysema, steroid dependent colitis; chronic kidney disease with an estimated glomerular filtration rate less than 30mg/mmol, venous thromboembolic disease with current treatment with vitamin K antagonist, Celiac disease, cirrhosis or steroid dependent arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Change in amount of vegetables eaten | Baseline, at 6 weeks, 10 weeks, 18 weeks and 30 weeks
  Self-reported number of vegetables eaten per day (e.g. 2 vegetables/day) will be obtained by the survey.
Change in weight (kg) | Baseline, at 6 weeks, 10 weeks, 18 weeks and 30 weeks
  Recorded from Electronic Medical Record (EMR) or weighed at weekly bag pick-up.
Change in Body mass index (kg/m^2) | Baseline, at 6 weeks, 10 weeks, 18 weeks and 30 weeks
  Recorded from EMR or calculated with height of record.

SECONDARY OUTCOMES:
Change in Glycosylated Hemoglobin level (percent of mmol/mol) | Baseline, at 6 weeks, 10 weeks, 18 weeks and 30 weeks
  Recorded from EMR.
Change in Blood pressure (mmHg) | Baseline, at 6 weeks, 10 weeks, 18 weeks and 30 weeks
  Recorded from EMR.

CONTACTS AND LOCATIONS:
Overall Officials: Donald RB Miles, MD, Principal Investigator — Johns Hopkins Community Physicians
Locations (1):
- Johns Hopkins Community Physicians at East Baltimore Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No